CLINICAL TRIAL: NCT02417636
Title: Impact of Task Shifting Type II for ART Delivery on Patient and Process Outcomes in Uganda
Brief Title: Sharing HIV/AIDS Responsibilities and Efforts
Acronym: SHARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Infectious Diseases Institute (Other)
Collaborators: Ministry of Health, Uganda (Other Government); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Infectious Diseases Institute, Principal Investigator, Makerere University
Organization: Makerere University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ST/0111/15
Record Dates: First submitted 2015-02-18; First posted 2015-04-15 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: PUBLIC HEALTH EVALUATION

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nurse-initiated and monitored ART (Experimental): This is an experimental task shifting of ART initiation and monitoring from a clinician-led model to a nurse-led model. Participants will be screened for eligibility for ART and the study and then enrolled initiated on ART by a Nursing Officers and then followed and monitored for ART adherence on a monthly basis for 12months. Quarterly, sexual behavior and quality of life questionnaires will be administered. CBC, CD4, HIV-1 Viral load, renal and liver function test will be done biannually. Nursing Officers will be free to consult with clinicians on the management of patients.
  Interventions: Other: Task Shifting
- Clinician - initiated and monitored ART (Active Comparator): This is Standard of Care for the Uganda Ministry of Health to compared with the experimental task shifting. Participants will be screened for eligibility for ART and the study and then enrolled initiated on ART by a Clinicians (Clinical Officer or Medical Officer) and then followed and monitored for ART adherence on a monthly basis for 12months. Quarterly, sexual behavior and quality of life questionnaires will be administered. CBC, CD4, HIV-1 Viral load, renal and liver function test will be done biannually.
  Interventions: Other: Task Shifting

INTERVENTIONS:
Other: Task Shifting — Participants will be screened for eligibility for ART and the study and then enrolled initiated on ART by a Nursing Officers and then followed and monitored for ART adherence on a monthly basis for 12months. Quarterly, sexual behavior and quality of life questionnaires will be administered. CBC, CD4, HIV-1 Viral load, renal and liver function test will be done biannually. Nursing Officers will be free to consult with clinicians on the management of patients.

SUMMARY:
PUBLIC HEALTH EVALUATION PROTOCOL on Impact of Task Shifting Type II for ART Delivery on Patient and Process Outcomes in Uganda

DETAILED DESCRIPTION:
SECTION 1: PROTOCOL SUMMARY Title: Impact of Task Shifting Type II for ART Delivery on Patient and Process Outcomes in Uganda Rationale: Health care worker shortages remain a major impediment to the scale-up of antiretroviral therapy (ART) in sub-Saharan Africa [1]. Sub-Saharan Africa suffers from the world's most pronounced crisis in human resources for health with 36 of 57 countries currently facing significant health worker shortages [2]. The health workforce crisis is further exacerbated by the HIV epidemic which thwarts efforts to expand and provide universal access to HIV/AIDS prevention, care and treatment. The shortage of health workers in sub-Saharan Africa presents a great challenge in service delivery, particularly in the scale up of antiretroviral therapy. According to the World Health Organization the global deficit of trained health care workers needed to provide essential health services in order to achieve the Millennium Development Goals, including the scaling up of biomedical interventions for HIV/AIDS is greater than 4 million [2]. In an attempt to meet the demand for ART services, the World Health Organization is coordinating a global effort to strengthen and expand the current health workforce and recommends task shifting as one potential strategy to meet the enormous demand for health care workers to provide HIV/AIDS care and treatment. This is particularly important at this time when patients are staying on ART for longer periods. Task shifting will allow physicians to see only severely ill patients thus freeing up their time for other duties. In addition, more patients can initiate ART because there are more available health workers to attend to them. There is however a need for empirical evidence to support the implementation of task shifting. For example, one critical question is whether candidate health worker cadres for task shifting of ART initiation and monitoring, will perform as well as doctors/clinicians. Country-specific evidence regarding this question is necessary for developing a task-shifting policy before initiating policy reforms in Uganda. Under PEPFAR funding a Public Health Evaluation (PHE) will be conducted in selected health facilities to determine the impact of implementing the WHO Global Recommendations and Guidelines on Task Shifting of HIV treatment from doctors and clinical officers to nurses.

Although task shifting for HIV treatment occurs de facto in several countries [3-10] , it is rarely institutionalized or allowed by national policies. Reliable data are necessary to better understand how and whether to include this strategy in national policy and operational guidelines.

The Investigators propose to conduct a randomized field intervention study to address the question of whether nurse-initiated and monitored ART is associated with inferior outcomes compared with clinician-initiated and maintained ART in treatment-naive, HIV positive individuals.

The findings of this study will contribute knowledge of how best to increase access to quality life-saving HIV treatment as well as improve health care worker skills and strengthen health system efficiency.

Primary Objectives:

To compare the following outcomes among HIV-infected individuals on antiretroviral therapy initiated and monitored by nurses and those initiated and monitored by clinicians at 6 and 12 months post ART initiation:

* virologic failure (≥ 1000 viral copies/ml)
* toxicity failure
* patient retention
* all-cause mortality

Secondary Objectives:

1. Compare immunological responses at time points 6 and 12 months post ART initiation
2. Compare accuracy of staging HIV-infected patients according to the WHO treatment guidelines as process outcomes among provider groups

Tertiary Objectives:

Test for HIV-1 drug resistance mutations (primary and secondary) among persons newly initiated on ART.

ELIGIBILITY:
Inclusion Criteria:

* Individuals will be eligible for the study if they:

  * are 18 years or older
  * have a confirmed HIV+ diagnosis at an accredited health facility according to the National HIV Testing Algorithm
  * are ART naive (except for short course mother-to-child transmission prophylaxis and post exposure prophylaxis not less than 6 months prior to study enrollment)
  * are clinically stable (no serious opportunistic infection, no other chronic condition)
  * are eligible for ART according to the Uganda National Treatment Guidelines

Exclusion Criteria:

* Individuals will not be eligible for the study if they

  * have more than grade 3 laboratory results for renal function, liver enzymes and hematology according to the National Institutes of Health Division of AIDS toxicity grading scale
  * are unwilling to give informed consent
  * anticipate moving from their current residence in the subsequent 24 months and
  * reside outside of a 40km radius (or more than 1 hour drive) of the selected study site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1760 (Actual)
Dates: Start 2015-02; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Treatment-limiting events that could occur on first-line ART | 12 months
  The primary study outcome is a composite endpoint of possible treatment-limiting events that could occur on first-line ART. These include virologic failure (viral load measure of ≥ 1000 copies/ml after 6 months of treatment), toxicity failure, loss to follow up and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bancroft, M.D., S.M., Principal Investigator — Centers for Disease Control and Prevention, Uganda
Locations (1):
- Mbale Regional Referral Hospital, Mbale, Uganda

REFERENCES:
- [Derived] Sekiziyivu BA, Bancroft E, Rodriguez EM, Sendagala S, Nasirumbi MP, Najjengo MS, Kiragga AN, Musaazi J, Musinguzi J, Sande E, Brad B, Dalal S, Byakika-Jayne T, Kambugu A. Task Shifting for Initiation and Monitoring of Antiretroviral Therapy for HIV-Infected Adults in Uganda: The SHARE Trial. J Acquir Immune Defic Syndr. 2021 Mar 1;86(3):e71-e79. doi: 10.1097/QAI.0000000000002567. PMID 33230029